CLINICAL TRIAL: NCT06066099
Title: A Controlled, Randomized, First-In-Human Study of AP31969 Investigating Single and Multiple Ascending Doses and the Effect of Food in Healthy Subjects
Brief Title: Single Ascending Dose, Multiple Ascending Dose, Food Effect Study With AP31969
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acesion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: AP31969-M101; 2023-505424-57-00 (Other: EU CT Number)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: Antiarrhythmic agent; Cardiac arrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Single Ascending Doses (Experimental): Participants will be randomized to receive a single oral dose of AP31969 or matching placebo in 1 of 5 groups.
  Participants in an additional food effect assessment group will be randomized to receive 2 single oral doses of AP31969 or matching placebo; 1 dose in fasted and 1 dose in fed state in a 2-period, fixed-sequence design (first fasted, then fed with at least 1 week washout between periods).
  Interventions: Drug: AP31969; Drug: Placebo
- Part B: Multiple Ascending Doses (Experimental): Participants will be randomized to receive multiple oral doses of AP31969 or matching placebo for 10 days in 1 of 4 groups.
  Interventions: Drug: AP31969; Drug: Placebo

INTERVENTIONS:
Drug: AP31969 — Oral tablets
Drug: Placebo — Oral tablets

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single doses (Part A) and multiple doses (Part B) of AP31969 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 18 years to 55 years, inclusive, at screening.
2. Weight: ≥50 kg, at screening.
3. Body mass index: 18.0 kg/m^2 to 30.0 kg/m^2, inclusive, at screening.
4. Sex : male or female; female participants may be of childbearing potential or of nonchildbearing potential (either surgically sterilized, physiologically incapable of becoming pregnant, or at least 1 year postmenopausal [amenorrhea duration of 12 consecutive months] and confirmed by a follicle-stimulating hormone test at screening).
5. In good physical and mental health on the basis of medical history, physical examination, clinical laboratory, 12-lead electrocardiogram (ECG), and vital signs, as judged by the Investigator.
6. Resting supine systolic blood pressure (BP) (average of 3 readings) between 140 and 90 mmHg (inclusive, at screening and [each] admission), and diastolic BP (average of 3 readings) between 90 and 50 mmHg (inclusive, at screening and [each] admission). If initial results do not meet these criteria, BP may be repeated if in the judgment of the Investigator there is a reason to believe the initial result is inaccurate (eg, white coat hypertension).
7. Computerized (12-lead) ECG recording without signs of clinically relevant pathology and with a QT-interval with Fridericia's correction (QTcF-interval) interval between 300 and 450 ms, inclusive, at screening and (each) admission.
8. Female participants must not be pregnant or lactating. Nonpregnancy will be confirmed for all female participants by a negative serum pregnancy test at screening and (each) admission.
9. Female participants of childbearing potential who have a fertile male sexual partner must agree to use highly effective contraception and not donate ova from 4 weeks prior to (the first) study drug administration until 90 days after the follow-up visit.
10. Male participants, if not surgically sterilized, who have a female sexual partner of childbearing potential must agree to use highly effective contraception and not donate sperm from (first) admission until 90 days after the follow-up visit.
11. Able to swallow up to 9 tablets of study drug (based on participant's own judgment after being informed about the possible number of tablets and the size of the tablets).
12. Willing and able to understand and comply with the protocol requirements, restrictions, and instructions listed in the informed consent form (ICF) and in the protocol and likely to complete the study as planned.
13. Willing and able to sign the ICF.

Exclusion Criteria:

1. Previous participation in the current study.
2. Employee of ICON or the Sponsor.
3. History of relevant drug and/or food allergies.
4. History of any illness or condition that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk when administering the study drug to the subject (with particular focus on cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, cerebrovascular, and neurological diseases including history of syncope and/or convulsions).
5. History of any major disorder capable of significantly altering the absorption, metabolism, or elimination of the study drug, constituting a risk when taking the study drug, or interfering with the interpretation of data in the opinion of the Investigator.
6. Personal or first-degree relative family history of congenital long QT syndrome or sudden death.
7. Presence of any signs of tremor in rest at screening or (at one of the) admission(s) to the clinical research center.
8. Use of any prescribed medication within 30 days prior to (first) admission, based on Investigator's judgment. An exception is made for hormonal contraceptives, which may be used throughout the study.
9. Use of any over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's wort) within 14 days prior to (first) admission, based on Investigator's judgment. An exception is made for acetaminophen/paracetamol, which is allowed up to 2 g/day.
10. Positive screen for hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus 1 and 2 antibodies, at screening. In case of vaccination against these diseases, inclusion is allowed.
11. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening or (at one of the) admission(s) to the clinical research center.
12. Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits).
13. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 2 years prior to screening.
14. Smoking on average more than 5 cigarettes, 1 cigar, or 1 pipe daily.
15. Participation in another drug study within 30 days prior to (the first) study drug administration in the current study, or in 4 or more drug studies within 12 months prior to (the first) study drug administration in the current study.
16. Donation or loss of more than 450 mL of blood within 60 days prior to (the first) study drug administration.
17. Significant and/or acute illness within 5 days prior to (the first) study drug administration that may impact safety assessments, in the opinion of the Investigator.
18. Unsuitable veins for blood sampling.
19. For the food effect group only: unwilling to consume high-fat, high-calorie meal.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experienced an Adverse Event | Up to a maximum of 48 days

SECONDARY OUTCOMES:
Parts A and B: Maximum Observed Plasma Concentration (Cmax) of AP31969 | Part A: Day 1 to Day 4; Part B: Day 1 to Day 12
Parts A and B: Time to Cmax (tmax) of AP31969 | Part A: Day 1 to Day 4; Part B: Day 1 to Day 12
Parts A and B: Terminal Elimination Half-life of AP31969 | Part A: Day 1 to Day 4; Part B: Day 1 to Day 12
Part A: Area Under the Plasma Concentration Time Curve (AUC) from Time 0 to Time of Last Quantifiable Concentration (AUC0-last) of AP31969 | Part A: Day 1 to Day 4
Part A: AUC from Time 0 Extrapolated to Infinity (AUC0-inf) of AP31969 | Part A: Day 1 to Day 4
Part B: AUC Over a Dosing Interval Tau (AUCtau) of AP31969 | Part B: Day 1 to Day 10
Part A: Apparent Clearance of AP31969 | Part A: Day 1 to Day 4
Part B: Apparent Clearance at Steady State of AP31969 | Part B: Day 1 to Day 10
Parts A and B: Apparent Volume of Distribution at Terminal Phase of AP31969 | Part A: Day 1 to Day 4; Part B: Day 1 to Day 10
Part B: Accumulation Ratio of AP31969 | Part B: Day 1 to Day 10
Parts A and B: Dose Normalized Cmax of AP31969 | Part A: Day 1 to Day 4; Part B: Day 1 to Day 10
Part A: Dose Normalized AUC0-last of AP31969 | Part A: Day 1 to Day 4
Part A: Dose Normalized AUC0-inf of AP31969 | Part A: Day 1 to Day 4
Part B: Dose Normalized AUCtau of AP31969 | Part B: Day 1 to Day 10
Part A: Food Effect on Cmax of AP31969 | Part A: Day 1 to Day 4 of fed and fasted treatment periods of the food effect assessment group
Part A: Food Effect on AUC0-last of AP31969 | Part A: Day 1 to Day 4 of fed and fasted treatment periods of the food effect assessment group
Part A: Food Effect on AUC0-inf of AP31969 | Part A: Day 1 to Day 4 of fed and fasted treatment periods of the food effect assessment group

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Operations, Study Director — Acesion Pharma
Locations (1):
- Acesion Pharma Investigational Site 10, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No